CLINICAL TRIAL: NCT05845073
Title: A Pilot Clinical Trial Assessing the Effect of Probiotic Supplementation on Antibiotic Associated Gastrointestinal Symptoms and Quality of Life
Brief Title: The Efficacy of a Probiotic for Antibiotic Associated Gastrointestinal Symptoms
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTB2022N104
Record Dates: First submitted 2023-03-27; First posted 2023-05-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: Probiotic; Antibiotic-associated Diarrhea; GI microbiome; Lactobacillus; Bifidobacterium
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Participants in this arm will receive a daily dose of 2x10^9 Colony Forming Units (CFU) of a multi strain probiotic (live bacterium), corresponding to 2 capsules twice daily, for the duration of antibiotic therapy, and 14 days thereafter.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants in this arm will receive an equivalent placebo for the duration of antibiotic therapy, and 14 day thereafter.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants in this arm will receive a daily dose of 2x10^9 Colony Forming Units (CFU) of a multi strain probiotic (live bacterium), corresponding to 2 capsules twice daily, for the duration of antibiotic therapy, and 14 days thereafter.
  Arms: Probiotic
Dietary Supplement: Placebo — Participants in this arm will receive an equivalent placebo for for the duration of antibiotic therapy, and 14 day thereafter.
  Arms: Placebo

SUMMARY:
This study evaluates the effect of a multistrain probiotic on gastrointestinal (GI) complaints and diarrhoea in subjects receiving short-term antibiotic (AB) treatment

DETAILED DESCRIPTION:
This study aims to investigate the safety and efficacy of live bacteria on gastrointestinal (GI) complaints and diarrhoea in subjects receiving short-term antibiotic (AB) treatment. The trial will be run in Germany and will recruit adult men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years and ≤65 years old
2. Body Mass Index 18.5-30 kg/m2
3. Generally in good health
4. Use of broad spectrum orally administered AB(s) for no more than 24h prior to V1 (penicillins, cephalosporins, quinolones, tetracyclines and lincomycins) for diagnosed infections other than those of GI, urinary or reproductive tract not requiring hospitalization, with a foreseen total duration of AB intake of 5-7 days
5. Having access to a smartphone/tablet or a computer with an internet access, and familiar with the use thereof (checked during the visit)
6. Readiness to keep dietary habits during the study
7. Readiness to avoid the use of any nutritional (e. g. prebiotic, probiotic), medical and further interventional options for management of GI complaints/diarrhoea (beyond the IP) during the study
8. Women of childbearing potential:

   * commitment to use contraception methods
   * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1

Exclusion Criteria:

1. More than 24h from the first dose of AB for diagnosed infections (as per inclusion criterion 4) until screening
2. Intravenously administered antibiotics
3. Taking AB in the last 30 days before starting current AB treatment
4. Taking any probiotic or prebiotic supplements in the last 30 days prior to screening
5. Using antidiarrheal medications / enemas on regular basis
6. Multimedication with microbiome-impacting medications within 30 days before enrolment (e.g. proton pump inhibitors antivirals/immunosuppressants, antidepressants)
7. Clinically relevant (as per investigator judgement) self-reported chronic diseases of GI tract (e.g. inflammatory bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease, diverticulitis, idiopathic esophageal reflux, malabsorption disorder, severe constipation), urinary tract, reproductive tract (e.g. endometriosis, adenomyosis, pelvic inflammatory disease, uterine fibroids) or metabolic (diabetes (type 1 or Type 2), familial hypercholestraemia, hereditary haemachromatosis) diseases
8. Any form of bowel preparation for endoscopy used in the last 3 months
9. Recent GI surgery (within the last 6 months)
10. Women of child-bearing potential: pregnancy, recently gave birth (within the last 6 months) and/or nursing
11. Recent Covid-19 infection (less than 4 weeks since the first negative SARS-CoV-2 (self) test after the infection)
12. Specific dietary restrictions (e.g. active phase of low Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols (FODMAP) diet)
13. Any dietary mode excluding passage of food via GI tract
14. High intake of alcohol (male subjects > 14 units per week, female subjects, >11 (1 unit corresponds to 360 mL beer, 45 mL spirits (40% alcohol) or 150 mL wine)
15. History of confirmed Clostridium difficile infection in the last 6 months
16. Known allergy or hypersensitivity to any ingredients of the IP
17. Previous adverse reactions to antibiotics
18. Artificial or damaged heart valves
19. History and/or presence of other clinically significant known (self-reported) condition/ disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

    * acute pancreatitis
    * immunodeficiency
    * eating disorder
    * recurrent diarrhoea
20. History of or current abuse of drugs or medication
21. Inability to comply with study requirements
22. Subjects who are deprived of their freedom by administrative or legal decision or who are in guardianship
23. Participation in another clinical study in the 30 days prior to V1 and during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Change in the Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) | Baseline (V1), Day 6 - 11 (V2)
  Change in Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome total score (max 78) from baseline (V1) to Day 6 - 11 (V2), where higher scores mean worse symptoms

SECONDARY OUTCOMES:
Difference in the Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) | Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) total score (max 78) between day 6 - 11 (V2) and day 20 - 25 (V3), where higher scores mean worse symptoms
Difference in the Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) | Baseline (V1), Day 20 - 25 (V3)
  Difference in Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) total score (max 78) from baseline (V1) to day 20 - 25 (V3) between intervention and placebo, where higher scores mean worse symptoms
Incidence of antibiotic-associated diarrhoea (AAD) | Through study completion, an expected average of 21 days
  Total incidence rate of antibiotic-associated diarrhoea (AAD) between intervention and placebo, defined as 2 or more days with a stool frequency of 3 or more a day and/or a stool consistency of 5 or more on the Bristol Stool Form Scale (BSFS), throughout the period between baseline (V1) and Day 20 - 25 (V3). The BSFS max score is 7, where lower scores indicate constipation and higher scores indicate diarrhoea
Duration of antibiotic associated diarrhoea (AAD) | Through study completion, an expected average of 21 days
  Difference in the average continuous days of antibiotic associated diarrhoea (defined as 2 or more days with a stool frequency of 3 or more a day and/or a stool consistency of 5 or more on the Bristol Stool Form Scale (BSFS)) in the intervention and placebo arms between baseline (V1) and day 20 - 25 (V3). The BSFS max score is 7, lower scores indicate constipation and higher scores indicate diarrhoea.
Difference in individual scores of Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) | Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in average individual Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome scores (max 7) from Day 6 - 11 (V2) to Day 20 - 25 (V3) where higher scores mean worse symptoms
Difference in individual scores of Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) | Baseline (V1), Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in average individual Gastrointestinal Symptom Rating Score - Irritable Bowel Syndrome (GSRS-IBS) scores (max 7) from Baseline (V1) to Day 6 - 11 (V2), and from Baseline (V1) to Day 20 - 25 (V3) where higher scores mean worse symptoms
Difference in Stool Consistency | Through study completion, an expected average of 21 days
  Difference in weekly stool consistency, as measured by the Bristol Stool Form Scale (BSFS) on a daily basis throughout the period between baseline (V1) and Day 20 - 25 (V3). BSFS max score 7 - lower scores indicate constipation, higher scores indicate diarrhea.
Difference in Stool Frequency | Through study completion, an expected average of 21 days
  Difference in weekly average stool frequency throughout the period between baseline (V1) and day 20 - 25 (V3).
Percentage with diarrhoea | Through study completion, an expected average of 21 days
  Percentage of participants who have developed diarrhoea (defined as proportion of subjects with stool classified on the Bristol Stool Form Scale (BSFS) as 5-7) throughout the period between baseline (V1) and day 20 - 25 (V3). BSFS max score is 7 - lower scores indicate constipation, higher scores indicate diarrhoea.
Duration of diarrhoea | Through study completion, an expected average of 21 days
  Duration of diarrhoea (defined as proportion of subjects with Bristol Stool Form Scale (BSFS) of 5-7/day) throughout the period between baseline (V1) and day 20 - 25 (V3). BSFS max score is 7 - lower scores indicate constipation, higher scores indicate diarrhoea.
Metabolomic Analysis of Faecal Samples | Baseline (V1), Day 6 - 11 (V2), Day 20 - 25 (V3)
  Targeted metabolomic analysis of faecal samples using liquid chromatography - mass spectrometry (LC-MS) for differences between baseline (V1), Day 6 - 11 (V2) and Day 20 - 25 (V3) including, but not restricted to succinate
Difference in Short Form 12 (SF-12) - Mental Component Score | Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Short Form-12 (SF-12) mental component score at Day 6 - 11 (V2) and Day 20 - 25 (V3). Higher scores indicate better mental health functioning (max score 100)
Difference in Short Form 12 (SF-12) - Physical Component Score | Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Short Form-12 (SF-12) physical component score at Day 6 - 11 (V2) and Day 20 - 25 (V3). Higher scores indicate better physical health (max score 100)
Difference in Short Form 12 (SF-12) - Mental Component Score (MCS) | Baseline (V1), Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Short Form-12 (SF-12) mental component score (MCS) from baseline (V1) to Day 6 - 11 (V2) and baseline (V1) to Day 20 - 25 (V3). Higher scores indicate better mental health (max score 100)
Difference in Short Form 12 (SF-12) - Physical Component Score (PCS) | Baseline (V1), Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Short Form-12 (SF-12) physical component score (PCS) from baseline (V1) to Day 6 - 11 (V2) and baseline (V1) to Day 20 - 25 (V3). Higher scores indicate better physical health (max score 100)

OTHER OUTCOMES:
Evaluation of Study Benefit | Day 20 - 25 (V3)
  Evaluation of benefit at study end by subject and the investigator (4 point scale, higher scores mean a better evaluation of the study product)
Matching records between blinded self-assessment | Day 20 - 25 (V3)
  Percentage of subject with matching records of blinded self-assessment concerning the IP type they received (verum, placebo) and the actual IP assignment
Stool Microbiome Assessment | Baseline (V1), Day 6 - 11 (V2), Day 20 - 25 (V3)
  Difference in Stool Microbiome analysis findings at baseline (V1), Day 6 - 11 (V2) and Day 20 - 25 (V3)
Change in body weight | Baseline (V1), Day 20 - 25 (V3)
  Change in body weight, measured in kilograms (Kg) between baseline (V1) and Day 20 - 25 (V3)

CONTACTS AND LOCATIONS:
Locations (1):
- analyze & realize GmbH, Berlin, Weißenseer Weg, Germany

IPD SHARING:
Plan to Share IPD: No